CLINICAL TRIAL: NCT04368000
Title: Prone Positioning in Awake Patients With COVID-19 Requiring Hospitalization
Acronym: PAPR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to lack of adherence to the protocol in the intervention arm.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Stacy Johnson, Associate Professor of Medicine, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00132123
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Respiratory Failure; COVID-19
Keywords: COVID-19; Respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Positioning (Experimental)
  Interventions: Behavioral: Intermittent prone positioning instructions
- Usual care (Active Comparator)
  Interventions: Behavioral: Usual care positioning with no instructions

INTERVENTIONS:
Behavioral: Intermittent prone positioning instructions — Participants will be given instructions to lie in the prone position for a duration of 1-2 hours, every 4 hours while awake.
  Arms: Prone Positioning
Behavioral: Usual care positioning with no instructions — Participants will not be given instructions to lie in the prone position for any duration.
  Arms: Usual care

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a major complication among patients with severe disease. In a report of 138 patients with COVID-19, 20% developed ARDS at a median of 8 days after the onset of symptoms, with 12.3% of patients requiring mechanical ventilation. Efficacious therapies are desperately needed. Supportive care combined with intermittent prone positioning may improve outcomes.

Prone positioning (PP) of patients with severe ARDS (when combined with other lung-protective ventilation strategies) is associated with a significant mortality benefit. In addition, PP for >12 hours in severe ARDS is strongly recommended by clinical practice guidelines. The aim of this study is to compare the outcomes of prone positioning versus usual care positioning in non-intubated patients hospitalized for COVID-19.

DETAILED DESCRIPTION:
In December 2019, an outbreak of a novel coronavirus (SARS-CoV-2) emerged in Wuhan, China and rapidly spread worldwide. The World Health Organization (WHO) declared the outbreak a pandemic on March 11th, 2020. The clinical disease (COVID-19) is mild in 81% of patients, severe disease occurs in 14%, and 5% of cases result in critical illness. The reported overall case fatality rate (CFR) is 2.3% in China, although the CFR varies widely (0.7- 7.2%) between regions. Older age is associate with increased mortality. The reported CFR is 8% among patients 70-79 years old and 15% in those 80 years and older.

Multiple therapies have been proposed based on in vitro evidence or anecdotal reports. Although, no high quality clinical trials have demonstrated an effective treatment regimen other than supportive care. Acute respiratory distress syndrome (ARDS) is a major complication among patients with severe disease. In a report of 138 patients with COVID-19, 20% developed ARDS at a median of 8 days after the onset of symptoms, with 12.3% of patients requiring mechanical ventilation. Efficacious therapies are desperately needed. Supportive care combined with intermittent prone positioning may improve outcomes.

Prone positioning (PP) of patients with severe ARDS (when combined with other lung-protective ventilation strategies) is associated with a significant mortality benefit. In addition, PP for >12 hours in severe ARDS is strongly recommended by clinical practice guidelines. Improvements in gas exchange, cardiac output, and clearance of secretions have been demonstrated with PP, and are thought to contribute to the survival benefits. Low quality evidence from case series and retrospective studies in awake, spontaneously breathing patients suggest PP is feasible, improves oxygenation, and may avoid the need for mechanical ventilation. A recent prospective observational study of early PP combined with high-flow nasal cannula or non-invasive mechanical ventilation was well tolerated and may help patients avoid intubation.

This study is a single-center non-blinded randomized controlled pragmatic feasibility study comparing the outcomes of prone positioning (intervention) versus usual care (control) in non-intubated patients hospitalized for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years)
* Suspected or Confirmed COVID-19 (Suspected: High clinical suspicion AND pending COVID-19 assay; Confirmed: Positive COVID-19 assay within 10 days)
* Scheduled for admission or already admitted to an inpatient hospital bed
* Patients must be enrolled within 48 hours of hospital admission

Exclusion Criteria:

* Pregnant
* Prisoner
* Contraindication to prone positioning: known increased intracranial pressure >30 mm Hg or cerebral perfusion pressure <60 mm Hg, increased abdominal pressure or risk for abdominal compartment syndrome, massive hemoptysis requiring urgent intervention, tracheal surgery or sternotomy during previous 14 days, facial surgery or serious facial trauma within 14 days, pacemaker implantation within 48 hours, unstable spine, femur, or pelvic fractures, chest tube, mean arterial pressure less than 65 mm Hg
* Lung transplant
* Burns on more than 20% of body surface
* Chronic respiratory failure requiring: mechanical ventilation via endotracheal device (e.g. tracheostomy tube, orotracheal tube, or nasotracheal tube)
* Inability to change position from supine to prone and prone to supine without assistance
* Receiving end of life care, comfort measures only, or hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Change in imputed partial pressure of oxygen over fraction of inspired oxygen (PaO2/FiO2) from peripheral capillary oxygen saturation over fraction of inspired oxygen (SpO2/FiO2) | 72 hours

SECONDARY OUTCOMES:
Change in imputed PaO2/FiO2 from SpO2/FiO2 | 48 hours
Proportion of participants requiring endotracheal intubation | Up to 8 weeks
Proportion of participants requiring mechanical ventilation | Up to 8 weeks
Proportion of participants transferred to intensive care for worsening respiratory failure | Up to 8 weeks
Proportion of participants who had escalated oxygen delivery needs | Up to 8 weeks
Average number of days hospitalized | Up to 8 weeks
Average number of ventilator-free days | Up to 8 weeks
Proportion of participants discharged from hospital on hospice | Up to 8 weeks
Proportion of participants with all-cause inpatient mortality | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stacy A Johnson, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No